CLINICAL TRIAL: NCT06177704
Title: Recurrent or Persistent Device Related Thrombus After Left Atrial Appendage Occlusion: The RE-DRT Study
Acronym: RE-DRT
Status: Not yet recruiting | Type: Observational
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal Investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Other Study IDs: RE-DRT
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Percutaneous Left Atrial Appendage Occlusion (LAAO); Device-related Thrombus (DRT); Thromboembolic Event; Major Cardioembolic Events; Major Bleeding - TIMI Classification
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diagnosis of probable/definite DRT after LAAO: Patients with diagnosis of probable/definite DRT after LAAO detected by transesophageal echocardiography (TEE) or cardiac computed tomography (CT).
  In all patients after the LAAO procedure, a first imaging evaluation at 45 to 90 days, and a second imaging evaluation at 12 months is recommended.
  In case of DRT diagnosis, and following the recent SCAI/HRS recommendations, a repeat imaging at 45- to 90-day intervals is recommended to assess for DRT resolution with eventual cessation of anticoagulation.
  In case of DRT resolution, a sequential imaging evaluation at ±90-day, ±180-day, and ±365 days after the imaging test where DRT was resolved is recommended

SUMMARY:
This study is a prospective, multicenter international trial aimed at assessing the actual incidence, identifying associated factors, and evaluating the clinical consequences of both persistent and recurrent device-related thrombus (DRT) following percutaneous left atrial appendage occlusion (LAAO).

While LAAO has shown efficacy in reducing the risk of stroke, device-related thrombus (DRT) remains a significant concern. The reported incidence of DRT varies, and it is associated with an elevated risk of ischemic stroke and death. The study highlights that persistent and recurrent DRT pose higher risks of thromboembolic events, and current data come from retrospective studies with non-standardized imaging follow-up protocols. The timing of imaging follow-up is crucial, and the study notes discrepancies in recommendations from expert statements. The EHRA/EAPCI suggests imaging at specific intervals post-procedure, while the SCAI/HRS recommends repeat imaging at shorter intervals to assess DRT resolution. The study underscores the need for dedicated prospective data to accurately determine the incidence, factors, and clinical impact of persistent and recurrent DRT after LAAO.

DETAILED DESCRIPTION:
BACKGROUND: Percutaneous left atrial appendage occlusion (LAAO) has emerged as a nonpharmacological alternative for stroke prevention in patients with non-valvular atrial fibrillation ineligible for chronic anticoagulation therapy. Large real-world observational studies have consistently reported the efficacy of LAAO in reducing the risk of ischemic stroke and systemic embolism, compared to predicted rates, without the need for anticoagulants. Despite ongoing refinement in LAAO procedural technique, significant challenges persist. Notably, device-related thrombus (DRT) remains the main concern after LAAO. The reported incidence rate varies, ranging from 3% to 7%, and has been associated with an elevated risk of ischemic stroke and all-cause death following LAAO. Several risk factors have been identified with DRT occurrence, most of which are non-modifiable. The diagnosis of DRT is followed by an intensification of the antithrombotic treatment. However, not all DRT are resolved, with a significant number persisting or recurring upon withdrawal of anticoagulation therapy. In these situations, the antithrombotic treatment must be maintained, increasing the risk of bleeding, and mitigating the potential benefits of LAAO.

Both persistent and recurrent DRT have been linked to an increased risk of thromboembolic events when compared to resolved DRT. In the pooled analysis of data from the PROTECT-AF and PREVAIL trials, around 12% of embolic events in patients with DRT occurred in the presence of multiple DRT episodes. The incidence of persistent DRT has been reported in one out of three patients diagnosed with DRT, with DRT recurrence occurring in one out of five patients. However, the real incidence of persistent and recurrent DRT is uncertain, as current data come from retrospective studies with non-standardized imaging follow-up protocols. This situation leads to a significant number of missed cases, increases the risk of bias, and likely underestimates the rate of persistent and recurrent DRT. The timing of the imaging follow-up can significantly affect the incidence of DRT. In consecutive patients examined through a pre-specified protocol, the incidence of specific findings would be much more accurate compared to imaging examinations based exclusively on a single adverse clinical event, where the real incidence and clinical associations cannot be accurately determined.

The EHRA/EAPCI expert LAAO statement recommends imaging within 6-24 weeks and then 12 months post-procedure, with no mention of imaging follow-up in case of persistent or recurrent DRT. In contrast, the recent SCAI/HRS expert consensus statement on transcatheter LAAO suggests that repeat imaging at 45- to 90-day intervals can be conducted to assess for DRT resolution and consider the eventual cessation of anticoagulation, although there is no evidence that support this recommendation. Finally, considering the substantial rate of recurrent DRT and its clinical implications, a long-term and sequential imaging follow-up strategy may be warranted. Therefore, there is an unmet need for dedicated prospective data to determine the real incidence, related factors, and clinical impact of persistent and recurrent DRT after LAAO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of probable/definite DRT after LAAO detected by transesophageal echocardiography (TEE) or cardiac computed tomography (CT).
* Age≥18 years old.

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing LAAO with a probable/definite diagnosis of DRT detected by transesophageal echocardiography (TEE) or cardiac computed tomography (CT).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic events (ischemic stroke, systemic embolism) | 1-month, 6-month, 1-year, 2-year
  Incidence of and thromboembolic events (ischemic stroke, systemic embolism) associated with persistent/recurrent DRT after LAAO

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ-UL, Québec, Quebec, Canada

REFERENCES:
- [Background] Mesnier J, Simard T, Jung RG, Lehenbauer KR, Piayda K, Pracon R, Jackson GG, Flores-Umanzor E, Faroux L, Korsholm K, Chun JKR, Chen S, Maarse M, Montrella K, Chaker Z, Spoon JN, Pastormerlo LE, Meincke F, Sawant AC, Moldovan CM, Qintar M, Aktas MK, Branca L, Radinovic A, Ram P, El-Zein RS, Flautt T, Ding WY, Sayegh B, Benito-Gonzalez T, Lee OH, Badejoko SO, Paitazoglou C, Karim N, Zaghloul AM, Agarwal H, Kaplan RM, Alli O, Ahmed A, Suradi HS, Knight BP, Alla VM, Panaich SS, Wong T, Bergmann MW, Chothia R, Kim JS, Perez de Prado A, Bazaz R, Gupta D, Valderrabano M, Sanchez CE, El Chami MF, Mazzone P, Adamo M, Ling F, Wang DD, O'Neill W, Wojakowski W, Pershad A, Berti S, Spoon DB, Kawsara A, Jabbour G, Boersma LVA, Schmidt B, Nielsen-Kudsk JE, Freixa X, Ellis CR, Fauchier L, Demkow M, Sievert H, Main ML, Hibbert B, Holmes DR Jr, Alkhouli M, Rodes-Cabau J. Persistent and Recurrent Device-Related Thrombus After Left Atrial Appendage Closure: Incidence, Predictors, and Outcomes. JACC Cardiovasc Interv. 2023 Nov 27;16(22):2722-2732. doi: 10.1016/j.jcin.2023.09.017. PMID 38030358
- [Background] Saw J, Holmes DR, Cavalcante JL, Freeman JV, Goldsweig AM, Kavinsky CJ, Moussa ID, Munger TM, Price MJ, Reisman M, Sherwood MW, Turi ZG, Wang DD, Whisenant BK. SCAI/HRS expert consensus statement on transcatheter left atrial appendage closure. Heart Rhythm. 2023 May;20(5):e1-e16. doi: 10.1016/j.hrthm.2023.01.007. Epub 2023 Mar 27. PMID 36990925
- [Background] Tzikas A, Holmes DR Jr, Gafoor S, Ruiz CE, Blomstrom-Lundqvist C, Diener HC, Cappato R, Kar S, Lee RJ, Byrne RA, Ibrahim R, Lakkireddy D, Soliman OI, Nabauer M, Schneider S, Brachmann J, Saver JL, Tiemann K, Sievert H, Camm AJ, Lewalter T. Percutaneous left atrial appendage occlusion: the Munich consensus document on definitions, endpoints, and data collection requirements for clinical studies. Europace. 2017 Jan;19(1):4-15. doi: 10.1093/europace/euw141. Epub 2016 Aug 18. PMID 27540038
- [Result] Holmes DR Jr, Korsholm K, Rodes-Cabau J, Saw J, Berti S, Alkhouli MA. Left atrial appendage occlusion. EuroIntervention. 2023 Feb 6;18(13):e1038-e1065. doi: 10.4244/EIJ-D-22-00627. PMID 36760206
- [Result] Holmes DR Jr, Reddy VY, Gordon NT, Delurgio D, Doshi SK, Desai AJ, Stone JE Jr, Kar S. Long-Term Safety and Efficacy in Continued Access Left Atrial Appendage Closure Registries. J Am Coll Cardiol. 2019 Dec 10;74(23):2878-2889. doi: 10.1016/j.jacc.2019.09.064. PMID 31806131
- [Result] Simard TJ, Hibbert B, Alkhouli MA, Abraham NS, Holmes DR Jr. Device-related thrombus following left atrial appendage occlusion. EuroIntervention. 2022 Jun 24;18(3):224-232. doi: 10.4244/EIJ-D-21-01010. PMID 35440430
- [Result] Alkhouli M, Alarouri H, Kramer A, Korsholm K, Collins J, De Backer O, Hatoum H, Nielsen-Kudsk JE. Device-Related Thrombus After Left Atrial Appendage Occlusion: Clinical Impact, Predictors, Classification, and Management. JACC Cardiovasc Interv. 2023 Nov 27;16(22):2695-2707. doi: 10.1016/j.jcin.2023.10.046. PMID 38030357
- [Result] Alkhouli M, Busu T, Shah K, Osman M, Alqahtani F, Raybuck B. Incidence and Clinical Impact of Device-Related Thrombus Following Percutaneous Left Atrial Appendage Occlusion: A Meta-Analysis. JACC Clin Electrophysiol. 2018 Dec;4(12):1629-1637. doi: 10.1016/j.jacep.2018.09.007. Epub 2018 Nov 1. PMID 30573129
- [Result] Mesnier J, Cepas-Guillen P, Freixa X, Flores-Umanzor E, Hoang Trinh K, O'Hara G, Rodes-Cabau J. Antithrombotic Management After Left Atrial Appendage Closure: Current Evidence and Future Perspectives. Circ Cardiovasc Interv. 2023 May;16(5):e012812. doi: 10.1161/CIRCINTERVENTIONS.122.012812. Epub 2023 May 16. PMID 37192309
- [Result] Asmarats L, Cruz-Gonzalez I, Nombela-Franco L, Arzamendi D, Peral V, Nietlispach F, Latib A, Maffeo D, Gonzalez-Ferreiro R, Rodriguez-Gabella T, Agudelo V, Alamar M, Ghenzi RA, Mangieri A, Bernier M, Rodes-Cabau J. Recurrence of Device-Related Thrombus After Percutaneous Left Atrial Appendage Closure. Circulation. 2019 Oct 22;140(17):1441-1443. doi: 10.1161/CIRCULATIONAHA.119.040860. Epub 2019 Oct 21. No abstract available. PMID 31634013
- [Result] Sedaghat A, Vij V, Al-Kassou B, Gloekler S, Galea R, Furholz M, Meier B, Valgimigli M, O'Hara G, Arzamendi D, Agudelo V, Asmarats L, Freixa X, Flores-Umanzor E, De Backer O, Sondergaard L, Nombela-Franco L, McInerney A, Korsholm K, Nielsen-Kudsk JE, Afzal S, Zeus T, Operhalski F, Schmidt B, Montalescot G, Guedeney P, Iriart X, Miton N, Saw J, Gilhofer T, Fauchier L, Veliqi E, Meincke F, Petri N, Nordbeck P, Rycerz S, Ognerubov D, Merkulov E, Cruz-Gonzalez I, Gonzalez-Ferreiro R, Bhatt DL, Laricchia A, Mangieri A, Omran H, Schrickel JW, Rodes-Cabau J, Nickenig G. Device-Related Thrombus After Left Atrial Appendage Closure: Data on Thrombus Characteristics, Treatment Strategies, and Clinical Outcomes From the EUROC-DRT-Registry. Circ Cardiovasc Interv. 2021 May;14(5):e010195. doi: 10.1161/CIRCINTERVENTIONS.120.010195. Epub 2021 May 18. PMID 34003661
- [Result] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Result] Glikson M, Wolff R, Hindricks G, Mandrola J, Camm AJ, Lip GYH, Fauchier L, Betts TR, Lewalter T, Saw J, Tzikas A, Sternik L, Nietlispach F, Berti S, Sievert H, Bertog S, Meier B; ESC Scientific Document Group. EHRA/EAPCI expert consensus statement on catheter-based left atrial appendage occlusion - an update. Europace. 2020 Feb 1;22(2):184. doi: 10.1093/europace/euz258. Epub 2019 Aug 31. No abstract available. PMID 31504441